CLINICAL TRIAL: NCT02084797
Title: Revisiting the Human Sweat Gland - Does Arginine Vasopressin Modulate Sweat Sodium Concentration Via the V2 Receptor?
Brief Title: V2 Receptor Effects on Fluid Regulation and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oakland University (Other)
Collaborators: Georgetown University (Other)
Responsible Party: Principal Investigator, Tamara Hew-Butler, Assoc Prof Exercise Science, Exercise Science, Oakland University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: RAM#4713
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Electrolyte Imbalance; Hyponatremia; Hypernatremia
Keywords: arginine vasopressin; sweat sodium; V2 antagonist; running
MeSH Terms: conditions — Hyponatremia; Hypernatremia; Diabetes Insipidus | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- all study participants (Experimental): All study participants received all interventions. V2R Antagonist: 30mg Tolvaptan tablet ingested 2 hours before exercise. V2R agonist: 0.2mg DDAVP tablet ingested 2 hours before exercise Placebo
  Interventions: Drug: V2R (Vasopressin 2 receptor)

INTERVENTIONS:
Drug: V2R (Vasopressin 2 receptor) — All ten subjects were used as their own controls in this double-blind, randomized controlled trial assessing the effect of the V2R on sweat sodium concentration via use of a V2R blocker (antagonist), stimulator (agonist), against a placebo (drug naive state).
  Other Names: V2R antagonist: tolvaptan (30mg tablet); V2R agonist: desmopressin (0.2mg tablet)

SUMMARY:
This primary aim of this study was to critically assess whether or not sweat water content and sodium concentration were acutely regulated by dynamic changes in antidiuretic hormone (arginine vasopressin or AVP) acting on the Vasopressin 2 receptor (V2R) during exercise. Secondary aims were to evaluate running performance and core temperature to further characterize the role of AVP in the coordinated balance of fluid and temperature homeostasis during exercise. The primary hypothesis was that activation of the V2R in sweat glands would result in water reabsorption and fluid conservation during endurance exercise.

DETAILED DESCRIPTION:
Ten healthy habitual runners (> 50km running per week) between 18-60 years of age participated in this double blind randomized control trial. Each subject presented to the exercise lab on four separate occasions. Trial 1 was a familiarization trial to determine each subject's maximal aerobic capacity and peak treadmill running speak (VO2 Peak test). Trials 2, 3 and 4 utilized the same exact protocol, differing only in pharmacological intervention. In a randomized, double-blind order (both participant and investigator blinded to the intervention), either a placebo pill, the V2 receptor antagonist tolvaptan (Samsca™, 30mg tablet), or the V2 receptor agonist desmopressin (DDAVP™, 0.2mg tablet) was ingested along with the CorTemp™ Core Temperature Sensor two hours before commencement of the Exercise Trial with 240mL of bottled water. The exercise protocol consisted of 60 minutes of treadmill running at 60% of peak speed (steady-state) followed by a performance test (the VO2 Peak test). Blood, saliva and urine, were collected before the exercise trial (baseline) and again after both the steady-state run and performance runs. Sweat was obtained from sweat patches after both the steady-state and performance runs. Core temperature, fluid intake, performance time, body weight, thirst and sodium palatability ratings were also assessed. Free access to water was allowed during the trial and all urine produced during the trial was measured and collected. The main outcome measure was sweat sodium concentration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (no acute or chronic medical conditions or regular prescription medication use), habitual (>50km/week)
* Distance runners between the ages of 18-60 years.

Exclusion Criteria:

* Individuals with chronic medical problems which require regular prescription medication
* Runners with pre-existing kidney problems
* Unable to sense thirst
* Difficulty swallowing
* Gastrointestinal disorders
* History of fainting associated with blood draw.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara D Hew-Butler, PhD, Principal Investigator — Oakland University; Joseph G Verbalis, MD, Study Director — Georgetown University
Locations (1):
- Oakland University, Rochester, Michigan, United States

REFERENCES:
- [Derived] Hew-Butler T, Hummel J, Rider BC, Verbalis JG. Characterization of the effects of the vasopressin V2 receptor on sweating, fluid balance, and performance during exercise. Am J Physiol Regul Integr Comp Physiol. 2014 Aug 15;307(4):R366-75. doi: 10.1152/ajpregu.00120.2014. Epub 2014 Jun 18. PMID 24944242

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received all three interventions in randomized fashion.
Groups:
- 1/Placebo, V2R Agonist, V2R Antagonist: This study was a double-blind randomized controlled trial in which all ten subjects participated in three trials under three separate pharmacological interventions: V2R antagonist, agonist and placebo conditions. A standardized exercise protocol was performed in the laboratory, separated by one week. Each subject served as his or her own control and the key which identified which intervention was utilized in the exact order (all tablets customized to appear identical) was unlocked only after data collection was completed. Therefore, all ten subjects participated in a total of thirty intervention exercise trials after the initial treadmill familiarization trial was completed.
  V2R (Vasopressin 2 receptor): All ten subjects were used as their own controls in this double-blind, randomized controlled trial assessing the effect of the V2R on sweat sodium concentration via use of a V2R blocker (antagonist), stimulator (agonist), against a placebo (drug naive state).
Period: Overall Study
Arm/Group | 1/Placebo, V2R Agonist, V2R Antagonist
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 1/Placebo, V2R Agonist, V2R Antagonist
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10
years of running experience [Mean (Standard Deviation); unit: years] | 8.8 (8.7)
BMI [Mean (Standard Deviation); unit: kg/m2] | 22.5 (3.3)
VO2 Peak [Mean (Standard Deviation); unit: ml/kg/minute] | 58.7 (6.2)
Peak treadmill running speed [Mean (Standard Deviation); unit: mph] | 11.0 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Sweat Sodium Concentration Obtained After the Steady-state Portion of the Trial
Description: Changes in sweat sodium concentration will parallel changes in urine sodium concentration with use of the V2R antagonist, agonist and placebo if the primary hypothesis is true (sweat sodium is regulated by the V2R, similar to how urine sodium is regulated by principle cells located within in the kidney collecting duct)
Time Frame: 4 study trials (4 weeks)
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | 1/Placebo, V2R Agonist, V2R Antagonist
Number analyzed (Participants) | 10
mEq/L
  Placebo | 80.1 (21.6)
  V2R Agonist | 76.8 (24.5)
  V2R Antagonist | 84.7 (25.7)

2. Secondary Outcome: Urine Sodium Concentration After the Steady-state Portion of the Trial
Description: Changes in urine sodium concentration after use of the V2R antagonist, agonist and placebo interventions will verify whether or not pharmacologic activation or inhibition was successfully induced.
Time Frame: 4 study trials (4 weeks)
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | 1/Placebo, V2R Agonist, V2R Antagonist
Number analyzed (Participants) | 10
mEq/L
  Placebo | 82.0 (48.5)
  V2R Agonist | 89.3 (21.5)
  V2R Antagonist | 16.4 (5.0)

3. Secondary Outcome: Blood Sodium Concentration
Description: Measurement of blood sodium concentration will determine if normonatremia (blood sodium concentrations within the normal physiological range of 135-145mmol/L) were maintained throughout the trial with appropriate fluid intake during the V2R antagonist, agonist and placebo intervention trials.
Time Frame: 4 study trials (4 weeks)
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | 1/Placebo, V2R Agonist, V2R Antagonist
Number analyzed (Participants) | 10
mEq/L
  Placebo | 143.6 (1.5)
  V2R Agonist | 144.3 (2.3)
  V2R Antagonist | 145.9 (2.0)

4. Secondary Outcome: Saliva Sodium Concentration
Description: Measurement of salivary sodium concentration will allow us to determine if the V2R antagonist, agonist and placebo interventions activate aquaporin-5 (AQP5) water channels that are also located in sweat glands. If the V2R acts on the sweat glands through AQP5, there should be parallel changes in sweat, urine and saliva sodium concentrations with each pharmaceutical intervention.
Time Frame: 4 trials (4 weeks)
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | 1/Placebo, V2R Agonist, V2R Antagonist
Number analyzed (Participants) | 10
mEq/L
  Placebo | 20.5 (11.0)
  V2R Agonist | 28.1 (9.5)
  V2R Antagonist | 31.0 (13.3)

5. Other Pre Specified Outcome: Body Weight
Description: Changes in body weight during the V2R antagonist, agonist and placebo conditions will provide researchers with an additional measure of overall fluid balance (fluid in versus fluid out) as well as an estimate of overall sweat water losses.
Time Frame: 4 trials (4 weeks)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Core Temperature
Description: Measurement of core temperature using an ingestible CorTemp sensor during the V2R antagonist, agonist and placebo trials will allow researchers to assess if fluid homeostasis and thermoregulation were intertwined in response to each pharmacological intervention.
Time Frame: 4 trials (4 weeks)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Thirst Rating
Description: To determine if fluid intake behaviors were appropriately regulated in response to the V2R antagonist, agonist and placebo conditions during exercise.
Time Frame: 4 trials (4 weeks)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Sodium Palatability Ratings
Description: To determine if sodium preference ratings were appropriately regulated in response to the V2R antagonist, agonist and placebo conditions during exercise.
Time Frame: 4 weeks (4 trials)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Performance
Description: To determine if exercise performance, as determined by overall exercise time, was affected in response to the V2R antagonist, agonist and placebo conditions.
Time Frame: 4 trials (4 weeks)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Fluid Intake
Description: as for outcome 7
Time Frame: 4 weeks (4 trials)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 1/Placebo, V2R Agonist, V2R Antagonist
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No